CLINICAL TRIAL: NCT02805803
Title: Quality of Life Assessment in Patients Undergoing Prolonged Suppressive Antibiotherapy for Prosthetic Joint Infection.
Acronym: PSA-QOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Principal Investigator, SMARMOR, Director, Groupe Hospitalier Diaconesses Croix Saint-Simon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ID RCB: 2015-A01702-47
Record Dates: First submitted 2016-06-15; First posted 2016-06-20 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Prosthetic Joint Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Quality of life questionary (Other): During this study of health and care procedure, we will assess the quality of life of patients treated with suppressive antibiotique therapy using three questionaries:
  * SF12
  * Beck
  * WOMAC
  Interventions: Other: Quality of life questionary

INTERVENTIONS:
Other: Quality of life questionary — Patients will be asked to fill out the questionaries before treatment initiation and at 3, 6 , 12 and 24 months after antibiotherapy initiation.
  Other Names: Depressive symptoms questionary; Joint functional questionary

SUMMARY:
Prosthetic joint infection (PJI) management is complex and requires prosthesis replacement when symptoms duration is greater than 30 days or debridement with modular set replacement when symptoms duration is lesser than one month. Nevertheless, the prolonged suppressive antibiotherapy (PSA) is the single treatment we can provide to high risk surgical patients and those who refuse reoperation.

There is limited data available on PSA modality, its tolerance and efficacy, this lack of data motivated us to concept a prospective study of long term patient follow up with PJI treated with prolonged suppressive antibiotherapy.

DETAILED DESCRIPTION:
Main objective:

Quality of life assessment of patients undergoing prolonged suppressive antibiotherapy for PJI.

Secondary objectives:

1. Depressive symptoms assessment in patients undergoing prolonged suppressive antibiotherapy for PJI.
2. Functional assessment in patients undergoing prolonged suppressive antibiotherapy for PJI.
3. Evaluation of PSA side effects
4. Evaluation of nutritional status
5. Evaluation of of PSA termination criteria

Methods:

The follow up oh this cohort will be conducted using 3 questionaries related to quality of life, joint stiffness and depressive symptoms.

Study type:

This is a study of health care procedure, evaluating the quality of life of patients undergoing prolonged suppressive antibiotherapy for PJI.

Sample size: all patients cared by our referral center of bone and joint infection, who meet protocol selection criteria will be included in the study, thus we are expecting to recruit 60 patients.

Study duration: 6 years.

Recruitment period: 4 years.

Maximal duration of data collection: 2 years.

Investigator center: Single center study.

Mean patient inclusion per year: 15 patients per year.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years old with hip or knee prosthetic infection who consented to participate in the study
* Non-eligible patient to surgical treatment
* Patient eligible to prolonged suppressive antibiotherapy

Exclusion Criteria:

* patient who does not meet eligibility criteria
* Patient living or traveling abroad for whom 2 years minimum follow up is impossible.
* Patient lawfully deprived of his liberty
* Patient not insured under social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11-09 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessment of patients undergoing prolonged suppressive antibiotherapy for PJI. | 2 years
  Method assessment : Short Form 12 questionary (SF12)

SECONDARY OUTCOMES:
1. Depressive symptoms assessment in patients undergoing prolonged suppressive antibiotherapy for PJI. | 2 years
  Method assessment : Beck depression inventory (BDI)
2. Functional assessment in patients undergoing prolonged suppressive antibiotherapy for PJI. | 2 years
  Method assessment : Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
3. Evaluation of PSA side effects | 2 years
  Method assessment : anamnesis and clinical examination
4. Evaluation of nutritional status | 2 years
  Method assessment : BMI and proteinuria measurement
5. Evaluation of PSA termination criteria | 2 years
  Monitoring :
  * Treatment failure in case of :
    * Side effects
    * Relapse of the infection
    * Persistance of the infection
  * The patient wishes terminate the treatment because of :
    * Side effects
    * The infection is controlled

CONTACTS AND LOCATIONS:
Overall Officials: Simon MARMOR, MD, Principal Investigator — Groupe Hospitalier Diaconesses Croix Saint-Simon
Locations (2):
- France (2):
  - Groupe Hospitalier Diaconesses Croix saint Simon, Paris
  - Groupe Hospitalier Dianconesses croix saint Simon, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No